CLINICAL TRIAL: NCT00480103
Title: Multi-Center Evaluation Program NCVD1H Intrauterine Embryo'S Development Assisted by ANECOVA ACVd1 Device
Brief Title: Intrauterine Embryo Development With ANECOVA Device
Acronym: ANECOVA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: INHERENT MODIFICATIONS NEEDED BEFORE PROCEEDING
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Collaborators: Anecova SA (Industry)
Responsible Party: Dr Carlos Simon, Instituto Valenciano de Infertilidad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NCVD1H
Record Dates: First submitted 2007-05-28; First posted 2007-05-30 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: Embryo morphological and chromosomal features; Implantation and pregnancy rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: in vivo (ANECOVA D-1) or in vitro culture in 25-µl droplets of cleavage medium (Medicult®) under paraffin oil

SUMMARY:
We aim to compare the morphological and chromosomal features of human embryos cultured In Vitro versus those developed in a new In Vivo culture system with encapsulation in utero as well as implantation and pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* Women age below 37
* Hormonal serum levels within normal ranges (FSH, LH, E2, PRL, P4, T4, TSH)
* Negative serologic screening for HIV, Hep B and C
* No uterine or ovarian alterations found by ultrasound
* Normal BMI (19 - 29 kg/m2).

Exclusion Criteria:

* At least 8 stage MII oocytes are not retrieved
* Endometriosis or PCO
* Severe male factor in the partner

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Velasco, Study Director — Affiliated
Locations (1):
- Instituto Valenciano de Infertilidad Spain, Valencia, Spain

REFERENCES:
- [Derived] Blockeel C, Mock P, Verheyen G, Bouche N, Le Goff P, Heyman Y, Wrenzycki C, Hoffmann K, Niemann H, Haentjens P, de Los Santos MJ, Fernandez-Sanchez M, Velasco M, Aebischer P, Devroey P, Simon C. An in vivo culture system for human embryos using an encapsulation technology: a pilot study. Hum Reprod. 2009 Apr;24(4):790-6. doi: 10.1093/humrep/dep005. Epub 2009 Mar 9. PMID 19273881